CLINICAL TRIAL: NCT00626457
Title: Promoting Healthy Weight With 'Stability Skills First' (Fresh Start Weight Loss Study)
Brief Title: Promoting Healthy Weight With 'Stability Skills First'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michaela Kiernan, Senior Research Scientist, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SU-02142008-1018; R01CA112594 (NIH)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance First (Experimental)
  Interventions: Behavioral: Behavioral weight-loss/lifestyle interventions
- Weight Loss First (Active Comparator)
  Interventions: Behavioral: Behavioral weight-loss/lifestyle interventions

INTERVENTIONS:
Behavioral: Behavioral weight-loss/lifestyle interventions — 6-month intervention (28 weekly classes)

SUMMARY:
Losing weight has many health benefits for women such as reducing the risk of heart attacks, high blood pressure, diabetes, and cancer. However, women often struggle with maintaining the weight they have lost. This may be because they need to learn skills for maintaining weight, not just losing weight.

When is the optimal time is to learn these maintenance skills? It may be better to lose weight first and then learn maintenance skills since people may feel good about the weight they have lost and be motivated to maintain. Alternatively, it may be better to learn maintenance skills first and then lose weight since they may experience how easy it is to use these maintenance skills and become confident they can maintain a weight loss in the future.

Therefore, this study will examine whether learning these maintenance skills--before or after losing weight--helps women succeed at maintaining weight loss.

DETAILED DESCRIPTION:
This randomized trial will test whether learning a novel set of 'stability skills' before losing weight improves long-term weight management (i.e., during a subsequent follow-up period once classes and staff contact have ended). Overweight/obese participants will be randomly assigned to one of two conditions (Maintenance First or Weight Loss First). In the Maintenance First condition, participants will learn stability skills during a novel 8-week maintenance program before participating in a standard 20-week behavioral weight-loss program. In the Weight Loss First condition (usual care/active comparator condition), participants will participate in a standard 20-week behavioral weight-loss program followed by a standard 8-week problem-solving skills maintenance program. Participants in both conditions will participate in identical standard 20-week behavioral weight-loss programs and be offered the same number of 90-minute weekly classes over the 6-month intervention period, (thus matching for time and attention from study-led health educators). Participants will be assessed at baseline and 6 months during the 6-month intervention period and at 12 and 18 months during the subsequent 12-month follow-up period (i.e., after classes and staff contact have ended). There will be no intervention staff contact during the 12-month follow-up, only 6, 12 and 18-month assessments. The primary aim will test whether participants in the Maintenance First condition gain less weight during the 12-month follow-up period (i.e., 6-18 months) than those in the Weight Loss First (active comparator) condition. Secondary questions of interest include examining psychometrics of lifestyle behavior questions (e.g., physical activity).

ELIGIBILITY:
Inclusion Criteria:

These criteria include: women of any ethnic background; age 21 years or older; BMI 27-40; non diabetic; not pregnant or not planning to become pregnant within the next year and a half; planning to remain in the area for the next year and a half; not following a special diet; not participating in any other research trial, not participating in another weight-loss program or weight or eating habits support group; able to participate in physical activity; free of heart disease, including stroke, heart attack, coronary artery bypass surgery, or balloon angioplasty; stable blood pressure, cholesterol, thyroid and/or hormone medications for at least 3 months; not taking weight-loss medications, and successful and timely completion of the eligibility process.

Exclusion Criteria:

These criteria include: all men; women younger than 21 years of age; BMI outside of range 27-40; diabetic; pregnant or planning to become pregnant within the next year and a half; not planning to remain in the area for the next year and a half; following a special diet; participating in another research trial; participating in another weight-loss program or weight or eating habits support group; not able to participate in physical activity; has a history of heart disease, including stroke, heart attack, coronary artery bypass surgery, or balloon angioplasty; taking blood pressure, cholesterol, thyroid, and/or hormone medications for less than 3 months; taking weight-loss medications, or unsuccessful and/or untimely completion of the eligibility process.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12-month follow-up period (6-18 months)
  Body weight will be measured at baseline, 6, 12, and 18 months on a California state-certified standard beam balance scale at the research center with participants in light clothing and without shoes.

SECONDARY OUTCOMES:
Change in physical activity | 6 months
  Physical activity will be assessed at baseline, 6, 12, and 18 months using the Stanford Leisure-Time Activity Categorical item (L-Cat). The L-Cat is self-administered and comprised of six ordered activity categories that range from inactive to very active. Participants pick the category that best describes their activity during the past month.
Pedometer steps | 6 months
  During the 6-month intervention sessions, participants will be asked to wear Omron dual axial pedometers (Model HJ-720ITC) every day during waking hours except when showering or swimming, and to record their steps per day and mean steps each week

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kiernan, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida, Gainesville, Florida

REFERENCES:
- [Result] Kiernan M, Moore SD, Schoffman DE, Lee K, King AC, Taylor CB, Kiernan NE, Perri MG. Social support for healthy behaviors: scale psychometrics and prediction of weight loss among women in a behavioral program. Obesity (Silver Spring). 2012 Apr;20(4):756-64. doi: 10.1038/oby.2011.293. Epub 2011 Oct 13. PMID 21996661
- [Result] Brown SD, Lee K, Schoffman DE, King AC, Crawley LM, Kiernan M. Minority recruitment into clinical trials: experimental findings and practical implications. Contemp Clin Trials. 2012 Jul;33(4):620-3. doi: 10.1016/j.cct.2012.03.003. Epub 2012 Mar 16. PMID 22449836
- [Result] Kiernan M, Brown SD, Schoffman DE, Lee K, King AC, Taylor CB, Schleicher NC, Perri MG. Promoting healthy weight with "stability skills first": a randomized trial. J Consult Clin Psychol. 2013 Apr;81(2):336-46. doi: 10.1037/a0030544. Epub 2012 Oct 29. PMID 23106759
- [Result] Kiernan M, Schoffman DE, Lee K, Brown SD, Fair JM, Perri MG, Haskell WL. The Stanford Leisure-Time Activity Categorical Item (L-Cat): a single categorical item sensitive to physical activity changes in overweight/obese women. Int J Obes (Lond). 2013 Dec;37(12):1597-602. doi: 10.1038/ijo.2013.36. Epub 2013 Apr 16. PMID 23588625